CLINICAL TRIAL: NCT03519451
Title: Use of a Smartphone Mobile Application (App) to Enhance Smoking Cessation Treatment - A Pilot Study
Brief Title: Use of a Smartphone Mobile Application (App) to Enhance Smoking Cessation Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-0720; NCI-2018-01158 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0720 (Other: M D Anderson Cancer Center); R43CA206682 (NIH)
Record Dates: First submitted 2018-04-26; First posted 2018-05-09 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Depression; Tobacco Use Disorder; Current Every Day Smoker
MeSH Terms: conditions — Depression; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group I (KickAsh smartphone mobile application) (Experimental): Participants receive KickAsh smartphone mobile application designed to help the learning of relaxation skills over 8 weeks.
  Interventions: Other: Internet-Based Intervention; Other: Questionnaire Administration
- Group II (Breathe2Relax smartphone mobile application) (Experimental): Participants receive Breathe2Relax smartphone mobile application designed to help improve mood and increase level of enjoyable activities over 8 weeks.
  Interventions: Other: Internet-Based Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Internet-Based Intervention — Given KickAsh smartphone mobile application
  Arms: Group I (KickAsh smartphone mobile application)
Other: Internet-Based Intervention — Given Breathe2Relax smartphone mobile application
  Arms: Group II (Breathe2Relax smartphone mobile application)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well smartphone mobile applications work in enhancing smoking cessation treatment in current smokers. Smartphone mobile applications may help current smokers quit smoking.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the acceptability and preliminary efficacy of a smartphone health application (app), Kick Ash, which will incorporate brief behavioral activation versus (vs.) a relaxation app, Breathe2Relax in a small randomized controlled trial of smokers with elevated depressive symptoms.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP I: Participants receive KickAsh smartphone mobile application designed to help the learning of relaxation skills over 8 weeks.

GROUP II: Participants receive Breathe2Relax smartphone mobile application designed to help improve mood and increase level of enjoyable activities over 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* MD Anderson patient between the ages of 18 to 65
* Current smoker (i.e., at least 1 cigarette or e-cigarette per day)
* Smoking for at least one year
* Willing to set a quit date in the next 30 days
* Not engaged in smoking cessation treatment other than the MDACC Tobacco Treatment Program
* Currently elevated depressive symptoms or a history of elevated depressive symptoms; (PHQ 2 = or > 1); current or past
* English speaking and ability to read and comprehend English
* Currently own an iOS mobile phone or tablet (iPhone; iPad) using iOS 9.0 or later and reports regular use (at least weekly) of at least 1 iOS app

Exclusion Criteria:

* Any medical or psychiatric condition, illness, disorder, or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator or Collaborator
* Subject considered by the investigator an unsuitable candidate for receipt of a smoking cessation treatment or unstable to be followed up throughout the entire duration of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-04-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
KickAsh group compliance with mood rating | Up to 8 weeks from start of study
  KickAsh group compliance with mood rating determined by questionnaires, phone calls, and interview.
KickAsh group change in activity level | Up to 8 weeks from start of study
  KickAsh group change in activity level determined by questionnaires, phone calls, and interview.
KickAsh group user satisfaction | Up to 8 weeks from start of study
  KickAsh group user satisfaction determined by questionnaires, phone calls, and interview.
Evidence of increased activity level in KickAsh and Breathe2Relax groups | Up to 8 weeks from start of study
  Increase in activity level determined by questionnaires, phone calls, and interview.
Evidence of improved mood in KickAsh and Breathe2Relax groups | Up to 8 weeks from start of study
  Evidence of improved mood determined by questionnaires, phone calls, and interview.
Evidence of greater smoking abstinence in KickAsh and Breathe2Relax groups | Up to 8 weeks from start of study
  Evidence of greater smoking abstinence determined by questionnaires, phone calls, and interview.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Minnix, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org